CLINICAL TRIAL: NCT00548002
Title: Combination Therapy With Fluoroquinolone in Staphylococcus Aureus Bacteremia
Acronym: FINLEVO
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Other Study IDs: 210275
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Staphylococcus Aureus; Bacteremia; Endocarditis; Sepsis
Keywords: Staphylococcus aureus; bacteremia; endocarditis; sepsis; fluoroquinolone; rifampin; levofloxacin; trovafloxacin
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia; Endocarditis; Sepsis | interventions — trovafloxacin; Levofloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 and 2: Patients were randomly assigned to receive either 1) standard treatment or 2) standard treatment combined with a fluoroquinolone (trovafloxacin or levofloxacin).
  Interventions: Drug: trovafloxacin and levofloxacin

INTERVENTIONS:
Drug: trovafloxacin and levofloxacin — Trovafloxacin: <60 kg 200 mg iv/orally once daily and >60 kg 300 mg iv/orally once daily Levofloxacin: < 60 kg 500 mg iv/orally once daily and >60 kg 500 mg iv/orally bid

SUMMARY:
To study whether fluoroquinolone (trovafloxacin or levofloxacin), added to standard treatment, could reduce the high mortality and complication rates in Staphylococcus aureus bacteremia.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with at least 1 blood culture positive for Staphylococcus aureus were included within 1 to 7 days of blood culture sampling.

Exclusion Criteria:

* age younger than 18 years
* imprisonment
* proven or suspected pregnancy
* breastfeeding, epilepsy
* another bacteremia during the previous 28 days
* polymicrobial bacteremia (_>3 microbes)
* history of allergy to any quinolone antibiotic
* previous tendinitis during fluoroquinolone therapy
* prior fluoroquinolone use for more than 5 days before randomization
* positive culture for Staphylococcus aureus only from a central intravenous catheter
* neutropenia (<0.5 x 109/L) or failure to supply an informed consent
* patients with bacteremia due to methicillin-resistant S. aureus and a S. aureus strain resistant to any fluoroquinolone
* patients with meningitis at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with at least 1 blood culture positive for Staphylococcus aureus were included within 1 to 7 days of blood culture sampling.
Enrollment: 430 (Actual)
Dates: Start 1999-01; Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Case fatality rate | At 28 days and at 3 months

SECONDARY OUTCOMES:
The number of complications (e.g. deep infections) observed after the first week antibiotic treatment, decrease in serum C-reactive protein concentration, length of antibiotic treatment, need for surgical intervention, and time to defervescence. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eeva Ruotsalainen, MD, Principal Investigator — Division of Infectious Diseases, Department of Medicine, Helsinki University Central Hospital, Helsinki, Finland
Locations (1):
- Division of Infectious Diseases, Department of Medicine, Helsinki University Central Hospital, Helsinki, HUS, Finland

REFERENCES:
- [Result] Ruotsalainen E, Jarvinen A, Koivula I, Kauma H, Rintala E, Lumio J, Kotilainen P, Vaara M, Nikoskelainen J, Valtonen V; Finlevo Study Group. Levofloxacin does not decrease mortality in Staphylococcus aureus bacteraemia when added to the standard treatment: a prospective and randomized clinical trial of 381 patients. J Intern Med. 2006 Feb;259(2):179-90. doi: 10.1111/j.1365-2796.2005.01598.x. PMID 16420547
- [Result] Ruotsalainen E, Sammalkorpi K, Laine J, Huotari K, Sarna S, Valtonen V, Jarvinen A. Clinical manifestations and outcome in Staphylococcus aureus endocarditis among injection drug users and nonaddicts: a prospective study of 74 patients. BMC Infect Dis. 2006 Sep 11;6:137. doi: 10.1186/1471-2334-6-137. PMID 16965625
- [Derived] Grumann D, Ruotsalainen E, Kolata J, Kuusela P, Jarvinen A, Kontinen VP, Broker BM, Holtfreter S. Characterization of infecting strains and superantigen-neutralizing antibodies in Staphylococcus aureus bacteremia. Clin Vaccine Immunol. 2011 Mar;18(3):487-93. doi: 10.1128/CVI.00329-10. Epub 2011 Jan 19. PMID 21248153